CLINICAL TRIAL: NCT01733836
Title: A Randomized Double Blind Placebo Controlled Single Institution Phase 2 Study of Metformin in Patients Undergoing Active Surveillance for Prostate Cancer.
Brief Title: Prostate Cancer Active Surveillance Metformin Trial
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: The reason for this decision is that this study is being merged with a larger multi-centre study using the same agent in the same population.
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MAS_001
Record Dates: First submitted 2012-11-20; First posted 2012-11-27 (Estimated); Last update posted 2013-05-24 (Estimated); Status verified 2013-05

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Metformin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Metformin (Experimental): 850mg BID
  Interventions: Drug: Metformin
- Placebo (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Metformin
  Arms: Metformin
Drug: placebo
  Arms: Placebo

SUMMARY:
To determine whether the use of metformin in patients with low-risk prostate cancer can delay progression to clinically significant prostate cancer.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to provide informed consent
* Men >= 18 years of age, and less than 80
* Men with biopsy proven, low-risk, localized prostate cancer (as defined below)
* Men choosing expectant management as primary treatment for prostate cancer
* Diagnostic biopsy performed within 4 months of screening visit
* Gleason score ≤ 6 in 3 cores or less with no Gleason pattern 4, less than 50% of any core involved in cancer
* Clinical stage T1c-T2a (Initial diagnosis of T1a/T1b obtained during a TURP is not allowed)
* Serum PSA ≤10 ng/mL
* Life expectancy greater than 5 years
* Normal kidney and hepatic function as defined by the following criteria:

  * Total bilirubin less than 1.5 X institutional upper limit of normal (ULN)
  * AST (SGOT)/ALT(SGPT) less than 1.5 X institutional ULN
  * Alkaline phosphatase less than 2 X institutional ULN
  * Creatinine less than 1.4 X institutional ULN
* Able to swallow and retain oral medication
* No exposure to metformin within 12 months of randomization
* No known hypersensitivity or intolerance to metformin hydrochloride
* No condition associated with increased risk of metformin hydrochloride-associated lactic acidosis (e.g., congestive heart failure defined as NYHA class III or IV function status, history of acidosis of any type, or habitual intake of ≥ 3 alcoholic beverages per day, or age greater than 80)
* English fluency allowing for patient reported outcomes completion

Exclusion Criteria:

* Any previous prostate cancer treatment (radiotherapy, chemotherapy, hormonal therapy, oral glucocorticoids, GnRH analogues)
* Diabetes including type 1 diabetes. Patients with known type 2 diabetes are eligible provided they have not been on metformin during the previous 12 months and are not on any other pharmacological agents.
* Concurrent or previous use of anabolic steroids or drugs with anti androgenic properties including 5-ARIs (dutasteride and finasteride)
* Prostate volume greater than 80 cc. (as per TRUS biopsy report)
* Prostatic surgery or procedure within 3 months of screening visit
* Severe BPH symptoms (IPSS ≥25, or ≥20 if already on α-blocker therapy)
* Other malignancies, with the exception of adequately treated nonmelanoma skin cancer, NMIBC or other solid tumors curatively treated with no evidence of disease for ≥ 5 years
* Planned or concurrent participation in other interventional randomized trials including exercise
* The presence of any other coexistent medical condition that in the opinion of the investigator would have the potential to significantly limit adherence to medication, or ability to absorb the medication including but not limited to psychiatric conditions, malabsorption syndromes or severe ischemic heart disease
* Known hypersensitivity or intolerance to metformin
* Concurrent or planned participation in randomized trials of weight loss or exercise interventions or trials targeting insulin, IGF-1 or their receptors, or PI3K inhibitors.

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-01; Primary Completion 2014-10 (Estimated); Study Completion 2014-10 (Estimated)

PRIMARY OUTCOMES:
Primary Clinical Outcome - Inhibition of Prostate Cancer | 18 months
  To assess the role of metformin on the inhibition of low-risk localized prostate cancer progression in men undergoing active surveillance for prostate cancer.
Primary Scientific Endpoint - ki67 index | 18 months
  To assess the effect of metformin on the cell cycle proliferation indices (ki67 index).

SECONDARY OUTCOMES:
Secondary Endpoint - Cell Cycle Proliferation (CCP) Score | 18 months
  To assess the effect of metformin on the cell cycle proliferation indices (CCP score)
Secondary Endpoint - Mechanism of Action | 18 months
  To assess the effect of metformin on systemic and local signalling axes and morphometric measurements relevant to its mechanism of action.
Secondary endpoint - Quality of Life | 18 months
  To assess the impact of metformin on Quality of Life (QoL) indices.
Secondary Endpoint - Prognostic Panel | 18 months
  To determine the utility of a prognostic panel of 31 cell cycle progression genes recently validated in prostate cancer.

CONTACTS AND LOCATIONS:
Locations (1):
- University Health Network, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Roy S, Malone S, Grimes S, Morgan SC. Impact of Concomitant Medications on Biochemical Outcome in Localised Prostate Cancer Treated with Radiotherapy and Androgen Deprivation Therapy. Clin Oncol (R Coll Radiol). 2021 Mar;33(3):181-190. doi: 10.1016/j.clon.2020.09.005. Epub 2020 Sep 29. PMID 32994091